CLINICAL TRIAL: NCT00176982
Title: Open Label Study of Hydroxychloroquine for Alopecia Areata, Alopecia Totalis
Brief Title: Plaquenil for Alopecia Areata, Alopecia Totalis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hordinsky, Maria K., MD (Individual)
Responsible Party: Maria Hordinsky MD, University of Minnesota
Organization: University of Minnesota (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0202M18141
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2009-08-13 (Estimated); Status verified 2009-08

CONDITIONS: Alopecia Areata
Keywords: treatment of alopecia areata
MeSH Terms: conditions — Alopecia Areata | interventions — Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine

SUMMARY:
Alopecia areata is an autoimmune condition resulting in hair loss and complete baldness (alopecia totalis). Published evidence says that it is mediated by T-lymphocytes. Plaquenil is an anti-inflammatory drug approved by the FDA for malaria, lupus erythematosus, and rheumatoid arthritis. It has an effect on T-lymphocyte mediated inflammation, making it a logical choice for a treatment trail for alopecia areata.

DETAILED DESCRIPTION:
Alopecia areata is a high prevalence autoimmune disease with significant consequences. Alopecia areata is a tissue restricted autoimmune disease directed at the hair follicle, resulting in hair loss. Patients frequently suffer severe psychiatric consequences. This is especially true of girls and young women who become bald. The incidence of alopecia areata in the USA (Minnesota is 20.2 per 100,000 person-years with a lifetime risk of approximately 1.7%. There is no significant gender difference. The disease is often chronic with a remitting, relapsing course. Although it responds to immunosuppression, generalized immunosuppression has significant morbidity and treatment is frequently frustrating and not successful. New treatment options are essential. With evidence that alopecia areata is a T-lymphocyte mediated autoimmune condition it has become a model system for the study of pathogenesis and treatment of T-cell mediated autoimmunity and as such is a model for a host of additional T-cell mediated autoimmune conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Severe alopecia areata: >75% loss of scalp hair or alopecia areata totalis: 100% loss of scalp hair above with or without loss of body hair (alopecia universalis) 2. Group I (8 subjects): Duration of disease less than 1 year 3. Group II (8 subjects): Duration of disease greater than 1 year 4. At least 18 years old 5. Able to give consent.

Exclusion Criteria:

1. Coexisting significant systemic disease that would increase risk of hydroxychloroquine (e.g. renal disease, liver disease, alcoholism, anemia, blood dyscrasia, psoriasis, porphyria) 2. Systemic immunosuppressive therapy within 3 weeks (e.g. prednisone, cyclosporin, azathioprine) 3. Immunosuppressive conditions (e.g. HIV infection, cancer immunotherapy genetic immunodeficiency 4. Medications with potential interaction to hydroxychloroquine (e.g. liver toxins, bone marrow toxins) 5. Pregnancy, or breast feeding 6. Women of child bearing potential not able or willing to use two methods of contraception at least one of which is not a hypersensitivity to 4-aminoquinolone compounds (chloroquine and hydroxychloroquine) 9. Glucose-6-phosphate deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16
Dates: Start 2002-04; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Percent hair regrowth in each quadrant of the scalp will be estimated and statistical analysis performed to determine if there was any significant regrowth compared to pre-treatment photographs.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Hordinsky, MD, Principal Investigator — University of Minnesota; Richard Kalish, MD, PhD, Principal Investigator — State Universiyt of New York at Stony Brook
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - State University of New York at Stony Brook, Stony Brook, New York